CLINICAL TRIAL: NCT03301766
Title: Adjunctive 5% Lidocaine Patches in the Treatment of Acute Non-radicular Low Back Pain in Patients Discharged From the Emergency Department
Brief Title: Adjunctive 5% Lidocaine Patches for Acute Non-radicular Low Back Pain in Emergency Department Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Delay for subject recruitment and then not feasible with COVID>
Sponsor: Cook County Health (Other Government)
Responsible Party: Principal Investigator, Neeraj Chhabra, Attending Physician, Department of Emergency Medicine, Principal Investigator, Cook County Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-510
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Low Back Pain
Keywords: lidocaine
MeSH Terms: conditions — Low Back Pain | interventions — Lidocaine; Transdermal Patch; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine 5% patch (Experimental): Patients will receive a 7 day supply (21 patches) of lidocaine 5% patches upon discharge from the emergency department in addition to "standard therapy" at the discretion of the treating emergency department physician.
  Interventions: Drug: lidocaine 5% patch; Drug: standard therapy
- Non-medicated patch (Active Comparator): Patients will receive a 7 day supply (21 patches) of non-medicated patches upon discharge from the emergency department in addition to "standard therapy" at the discretion of the treating emergency department physician.
  Interventions: Drug: standard therapy; Drug: Non-medicated patch

INTERVENTIONS:
Drug: lidocaine 5% patch — transdermal patch
  Arms: Lidocaine 5% patch
Drug: standard therapy — Drugs prescribed at the discretion of the treating physician (acetaminophen, NSAIDs, muscle relaxants, etc)
Drug: Non-medicated patch — non-medicated patch
  Arms: Non-medicated patch

SUMMARY:
This study will evaluate the addition of lidocaine % transdermal patches to standard therapy in the treatment of acute non-radicular low back pain in patients discharged from the Emergency Department. In addition to standard therapy, half of the participants will receive medicated patches while the other half will receive non-medicated patches.

DETAILED DESCRIPTION:
Low back pain is a common emergency department (ED) chief complaint. Multiple therapies have been evaluated in the treatment of ED patients with low back pain including acetaminophen, NSAIDS, opioids, steroids, and muscle relaxants.

Lidocaine is a local anesthetic that can be administered by various routes. It is used in a transdermal patch for the treatment of pain. It is commonly used for focal causes of pain, including low back pain. The addition of lidocaine 5% patches to standard low back pain therapy has not been rigorously evaluated, although it is frequently used.

ELIGIBILITY:
Inclusion Criteria:

* pain originating between the lower border of the scapulae and the upper gluteal folds
* treating ED physician plan for discharge of the patient

Exclusion Criteria:

* radicular pain defined as pain radiating below the gluteal folds
* direct trauma to the back within previous month
* pain of greater than 2 weeks duration or greater than 1 LBP episode per month in the past 3 months
* patient being pregnant or lactating; no access to phone or ability to participate in follow-up phone calls
* known allergy to lidocaine or skin breakdown over site of pain
* treating physician plan for opioid prescription (tramadol, codeine, hydrocodone)
* personal history of malignancy, fever (temperature greater than 37.9ºC), or previous spinal surgery
* patients who are detainees
* previous enrollment in the study

Ages: 24 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NRS) | 1 week
  Patient description of pain on a scale of 0-10

SECONDARY OUTCOMES:
Roland-Morris-24 back pain disability scale | 1 week and 1 month
  24 point back pain disability scale
Numerical Pain Rating Scale (NRS) | 1 month
  Patient description of pain on a scale of 0-10

OTHER OUTCOMES:
Repeat visits | 1 week and 1 month
  Repeat visits to an emergency department

CONTACTS AND LOCATIONS:
Locations (1):
- John H Stroger Jr Hospital of Cook County, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No